CLINICAL TRIAL: NCT04520321
Title: A Phase 1/ Phase 2 Study Evaluating the Safety and Efficacy of the Investigational New Drug TTHX1114(NM141) on the Regeneration of Corneal Endothelial Cells in Patients With Corneal Endothelial Dystrophies Following Intracameral Delivery
Brief Title: A Phase 1/ Phase 2 Study of TTHX1114(NM141)
Acronym: INTREPID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Trefoil Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTHX-001
Record Dates: First submitted 2020-08-14; First posted 2020-08-20 (Actual); Results first posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2022-10

CONDITIONS: Corneal Endothelial Dystrophy; Fuchs Endothelial Corneal Dystrophy; Pseudophakic Bullous Keratopathy; Endothelial Dysfunction
MeSH Terms: conditions — Corneal Dystrophy, Posterior Polymorphous, 1; Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Intervention Model Description: Randomized, Masked, Vehicle-controlled, Dose-escalation study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Vehicle (placebo) (Placebo Comparator): Placebo weekly x 4
  Interventions: Other: Vehicle (placebo)
- Low dose (Experimental): TTHX1114(NM141) low-dose weekly x 4
  Interventions: Drug: TTHX1114(NM141)
- Mid-dose (Experimental): TTHX1114(NM141) mid-dose weekly x 4
  Interventions: Drug: TTHX1114(NM141)
- High-dose (Experimental): TTHX1114(NM141) high-dose weekly x 4
  Interventions: Drug: TTHX1114(NM141)

INTERVENTIONS:
Drug: TTHX1114(NM141) — engineered FGF-1 delivered intracamerally
  Arms: High-dose; Low dose; Mid-dose
Other: Vehicle (placebo) — Placebo
  Arms: Vehicle (placebo)

SUMMARY:
Prospective, multicenter, randomized, masked, vehicle-controlled, dose-escalation study

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, masked, vehicle-controlled, dose-escalation study that will include an observational (no intervention) sub-study. Eligible subjects with moderate to severe corneal endothelial dystrophy (defined as Endothelial Cell Density < 2000 mm^2) in at least one eye will be enrolled and randomized.

ELIGIBILITY:
Key Inclusion Criteria:

* Fuchs Endothelial Corneal Dystrophy, pseudophakic bullous keratopathy, or endothelial dysfunction/ insufficiency due to surgical intervention diagnosed more than 6 months prior to Study Day 0
* Central endothelial cell count of < 2000 mm^2 in at least one eye as determined by the central reading facility

Key Exclusion Criteria:

* Conditions that would impair examination of the anterior chamber structure
* Documented repeated elevated intra ocular pressure (in either eye)
* Corneal transplant (in either eye)
* Posterior Polymorphous Corneal Dystrophy (PPCD)
* History of uveitis or herpetic keratitis
* Cataract surgery within the past 3 months
* Refractive surgery (in the Study Eye)
* Anterior Chamber IOL placement (in the Study Eye)
* Active extra-ocular inflammation from any non-infectious or infectious cause within the past 6 months
* Expected or planned ocular surgery within the next 3 months
* Use of cytotoxic chemotherapy within the last 1 month
* Treatment with a rho kinase inhibitor within the last 3 months
* Use of cyclosporine ophthalmic emulsion or lifitegrast ophthalmic solution in the last 30 days
* Systemic or ophthalmic corticosteroid use in the 30 days prior to Study Day 0 unless approved by the Medical Monitor
* History of significant allergy, hypersensitivity, or intolerance to any drug compound, food, or other substance
* Unwilling to use birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Tremblay, RN BSN, Study Director — Trefoil Therapeutics
Locations (8):
- United States (8):
  - North Bay Eye Associates, Inc., Petaluma, California
  - Levenson Eye Associates, Inc, Jacksonville, Florida
  - Chicago Corneal Consultants, Hoffman Estates, Illinois
  - Price Vision Group, Indianapolis, Indiana
  - Tauber Eye Center, Kansas City, Missouri
  - Vance Thompson Vision - Omaha, Omaha, Nebraska
  - Alterman, Modi and Wolter, Poughkeepsie, New York
  - Vance Thompson Vision - Sioux Falls, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vehicle (Placebo) | Low Dose | Mid-dose | High-dose
Started | 5 | 7 | 3 | 7
Completed | 5 | 7 | 3 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle (Placebo) | Low Dose | Mid-dose | High-dose | Total
Number analyzed (Participants) | 5 | 7 | 3 | 7 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.6 (11.8) | 75.7 (7.8) | 81.3 (11.0) | 68.9 (11.1) | 74.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 2 | 7 | 19
  Male | 0 | 2 | 1 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 7 | 3 | 7 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 7 | 3 | 7 | 22
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: DLTs/ Adverse Reactions
Description: Suspected Adverse Reactions Reported Following Study Drug Adminsitration
Time Frame: Day 90
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle (Placebo) | Low Dose | Mid-dose | High-dose
Number analyzed (Participants) | 5 | 7 | 3 | 7
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Vehicle (Placebo) | Low Dose | Mid-dose | High-dose
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/7 | 0/3 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7 | 0/3 | 0/7
Other Adverse Events (participants affected / at risk) | 2/5 | 1/7 | 2/3 | 3/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (Placebo) (N=5) | Low Dose (N=7) | Mid-dose (N=3) | High-dose (N=7)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 (0) | 0 | 1 | 1
Foreign body sensation in eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iritis (Eye disorders) | 0 (0) | 0 | 0 | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 | 0 | 1
Punctate keratitis (Eye disorders) | 0 (0) | 0 | 0 | 1
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 1 (1) | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT04520321/Prot_001.pdf